CLINICAL TRIAL: NCT02815254
Title: The Effect of Exercise in Elderly Hip Fracture Patients: a Clinical Randomised Trial
Brief Title: Better Hips- Better Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Braseth rehabilitation centre (Unknown)
Responsible Party: Principal Investigator, Astrid Bergland, Professor, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1441
Record Dates: First submitted 2015-04-21; First posted 2016-06-28 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Hip Fracture
Keywords: Physiotherapy; hip fracture; rehabilitation; high dose exercise; low dose exercise
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose exercise intervention (Active Comparator)
  Interventions: Other: Low intensity functional exercise
- High dose exercise intervention (Experimental)
  Interventions: Other: High intensity functional exercise

INTERVENTIONS:
Other: High intensity functional exercise
  Arms: High dose exercise intervention
Other: Low intensity functional exercise
  Arms: Low dose exercise intervention

SUMMARY:
The focus of this project are elderly people who have experienced hip fracture and need at least two weeks rehabilitation after discharge from hospital. The aim is to increase the evidence-based knowledge base for planning and appropriate follow-up intervention for patients with hip fracture on short-term / rehabilitation stays. In this study the investigators want to explore whether training High Intensity Functional Exercises (HIFE) , of short duration ie a 2- 4 week program and frequent intervention ie 5 times per week has a significant positive effect on physical function, pain and quality of life. The main aim is to explore whether a high intensive strength and balance training program has better effect than a low intensive strength and balance training program on functional status measured by Short Physical Performance Battery (SPPB) in patients with hip fractures. Another aims is to explore whether this high intensive strength and balance training program has better effect than a 'low intensive strength and balance training program' on pain, endurance and quality of life measured respectively Numeric Pain Rating Scale (NPR), 6-minute walk test and SF-36. The study is a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Fractura colli femoris, pertrochantar or subtrochantar)
* Discharged from hospital within 3 weeks since surgery.
* Need of minimum two weeks rehabilitation
* Life expectancy of more than one month
* Able to walk at least 3 m with walking aid
* Willingness to participate
* Able to follow instructions
* 65 years or older

Exclusion Criteria:

-Other reasons for gait impairment than hip fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-11; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
The Short Physical Performance Battery | November 2015 -October 2018 (up to 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Bergland, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Braseth rehabilitation centre, Røyken, Norway

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134